CLINICAL TRIAL: NCT04059172
Title: Efficacy of Combined Ibuprofen and Acetaminophen Therapy Versus Ibuprofen Alone Versus Placebo Alone for Pain of Initial Orthodontic Wire Insertion: a Randomized Controlled Trial
Brief Title: Efficacy of Combined Ibuprofen and Acetaminophen Therapy Versus Ibuprofen Alone Versus Placebo Alone for Pain Management
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1449
Record Dates: First submitted 2019-08-07; First posted 2019-08-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pain, Orofacial
MeSH Terms: conditions — Facial Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Two investigational groups and a placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Ibuprofen, acetaminophen and placebo tablets have been prepared to look identical by a pharmacy. The appropriate tablets are placed in a blister pack to be delivered to the study participant. The number of tablets are the same for each blister in all blister packs.
  The study participant, care provider, investigators and the outcomes assessor are all blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ibuprofen (Active Comparator): one 200 mg tablet of ibuprofen and 2 placebo tablets
  Interventions: Drug: Ibuprofen 200 mg
- Ibuprofen and acetaminophen (Experimental): one 200 mg table of ibuprofen and two 325 mg tablets of acetaminophen
  Interventions: Drug: Ibuprofen 200 mg and acetaminphen 650 mg
- Placebo (Placebo Comparator): 3 tablets of tableting compounds with no active ingredients
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ibuprofen 200 mg and acetaminphen 650 mg — For morning appliance placement: dose #1 at approximately 9:00 a.m. as appointment starts; dose #2 6 hours later (3:00 p.m- or as soon after school and close to 3 pm as possible.); dose #3 another 6 hours later (9:00 p.m.); dose #4 the following morning upon waking (approximately 24 hours from start and patient will record the time), doses #5 through #7 will be taken every morning upon waking on the second, third, and fourth days, respectively.
  For afternoon appliance placement: dose #1 at approximately 2:00 p.m. as appointment starts; dose #2 6 hours later (8:00 p.m.); dose #3 the following morning upon waking (approximately 12 hours later and patient will record the time); dose #4 6 hours later from dose #3 (approximately 24 hours from the initial dose) around 2:00 p.m. (or as soon after school as possible) doses #5 through #7 will be taken every afternoon at 2:00 p.m. on the second, third, and fourth days, respectively.
  Arms: Ibuprofen and acetaminophen
Drug: Ibuprofen 200 mg — For morning appliance placement: dose #1 at approximately 9:00 a.m. as appointment starts; dose #2 6 hours later (3:00 p.m- or as soon after school and close to 3 pm as possible.); dose #3 another 6 hours later (9:00 p.m.); dose #4 the following morning upon waking (approximately 24 hours from start and patient will record the time), doses #5 through #7 will be taken every morning upon waking on the second, third, and fourth days, respectively.
  For afternoon appliance placement: dose #1 at approximately 2:00 p.m. as appointment starts; dose #2 6 hours later (8:00 p.m.); dose #3 the following morning upon waking (approximately 12 hours later and patient will record the time); dose #4 6 hours later from dose #3 (approximately 24 hours from the initial dose) around 2:00 p.m. (or as soon after school as possible) doses #5 through #7 will be taken every afternoon at 2:00 p.m. on the second, third, and fourth days, respectively.
  Arms: Ibuprofen
Drug: Placebo oral tablet — For morning appliance placement: dose #1 at approximately 9:00 a.m. as appointment starts; dose #2 6 hours later (3:00 p.m- or as soon after school and close to 3 pm as possible.); dose #3 another 6 hours later (9:00 p.m.); dose #4 the following morning upon waking (approximately 24 hours from start and patient will record the time), doses #5 through #7 will be taken every morning upon waking on the second, third, and fourth days, respectively.
  For afternoon appliance placement: dose #1 at approximately 2:00 p.m. as appointment starts; dose #2 6 hours later (8:00 p.m.); dose #3 the following morning upon waking (approximately 12 hours later and patient will record the time); dose #4 6 hours later from dose #3 (approximately 24 hours from the initial dose) around 2:00 p.m. (or as soon after school as possible) doses #5 through #7 will be taken every afternoon at 2:00 p.m. on the second, third, and fourth days, respectively.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of a combined ibuprofen and acetaminophen regimen in controlling discomfort for 4 days after initial orthodontic appliance placement as compared to ibuprofen alone or a placebo. The hypothesis is that combined ibuprofen and acetaminophen therapy will effectively provide better pain control than ibuprofen alone or a placebo after orthodontic appliance placement.

DETAILED DESCRIPTION:
Orthodontic pain is often reported for the first 4 days after the appliances are attached. This study will investigate two modes of pain management versus a placebo. Consented subjects will be randomly assigned to one of 3 groups: Group A, a combined and simultaneous therapy of 200 mg ibuprofen and 650 mg acetaminophen (3 pills total) taken orally at set time intervals (0 h, 6 h, 12 h, and 24h, 48h, 72h, and 96h); Group B, ibuprofen alone (200 mg) taken orally at same time intervals (1 ibuprofen and 2 placebo pills); Group C, placebo taken orally at the same time intervals (3 placebo pills).

The study will be blinded for the investigators, patients, and statisticians.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to begin comprehensive orthodontic treatment (banding/bonding of at least 10 teeth in 1 arch and archwire placement in at least 1 arch);
* extractions, if required, performed at least 2 weeks before appliance and archwire placement;
* healthy with no significant medical findings;
* no prophylactic antibiotic coverage required;
* currently not taking antibiotics or analgesics;
* no contraindications to the use of acetaminophen or ibuprofen; and
* minimum age of 12 years

Exclusion Criteria:

* Under the age of 12 or over the age of 80,
* prisoners,
* pregnant women,
* decisionally challenged individuals,
* allergy to either medication,
* history of kidney disease,
* liver damage or disease,
* alcoholism/use of 3 or more alcoholic drinks during study period,
* use of blood thinners,
* stomach ulcers or
* stomach bleeding.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in visual analogue score (VAS) over time | 0 hours, 6 hours, 12 hours, and 24 hours, 48 hours, 72 hours, and 96 hours after placement of appliances
  Primary outcomes with be the pain values recorded by subjects when chewing on the 100-mm VAS at set times.The VAS line for each time period will be 100 mm long with no intermediate delineations. Each end will be marked with "no pain" on the left, and "worst possible pain" on the right.

SECONDARY OUTCOMES:
Dosing Compliance | to be recorded at 0 hours, 6 hours, 12 hours, and 24 hours, 48 hours, 72 hours, and 96 hours after placement of appliances.
  The VAS containing booklet will ask the patient to record if he or she took all of the pills provided at each time point to monitor compliance. Additionally, the VAS containing booklet will ask the patient to record will ask if any additional medication was taken and if so, to name the additional medication and dosage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, School of Dental Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers.

REFERENCES:
- [Background] Angelopoulou MV, Vlachou V, Halazonetis DJ. Pharmacological management of pain during orthodontic treatment: a meta-analysis. Orthod Craniofac Res. 2012 May;15(2):71-83. doi: 10.1111/j.1601-6343.2012.01542.x. PMID 22515183
- [Background] Bartzela T, Turp JC, Motschall E, Maltha JC. Medication effects on the rate of orthodontic tooth movement: a systematic literature review. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):16-26. doi: 10.1016/j.ajodo.2008.08.016. PMID 19121496
- [Background] Bernhardt MK, Southard KA, Batterson KD, Logan HL, Baker KA, Jakobsen JR. The effect of preemptive and/or postoperative ibuprofen therapy for orthodontic pain. Am J Orthod Dentofacial Orthop. 2001 Jul;120(1):20-7. doi: 10.1067/mod.2001.115616. PMID 11455373
- [Background] Doll GM, Zentner A, Klages U, Sergl HG. Relationship between patient discomfort, appliance acceptance and compliance in orthodontic therapy. J Orofac Orthop. 2000;61(6):398-413. doi: 10.1007/pl00001908. English, German. PMID 11126015
- [Background] Hyllested M, Jones S, Pedersen JL, Kehlet H. Comparative effect of paracetamol, NSAIDs or their combination in postoperative pain management: a qualitative review. Br J Anaesth. 2002 Feb;88(2):199-214. doi: 10.1093/bja/88.2.199. PMID 11878654
- [Background] Romsing J, Moiniche S, Dahl JB. Rectal and parenteral paracetamol, and paracetamol in combination with NSAIDs, for postoperative analgesia. Br J Anaesth. 2002 Feb;88(2):215-26. doi: 10.1093/bja/88.2.215. PMID 11878655
- [Background] Jones ML, Chan C. Pain in the early stages of orthodontic treatment. J Clin Orthod. 1992 May;26(5):311-3. No abstract available. PMID 1430181
- [Background] Jones M, Chan C. The pain and discomfort experienced during orthodontic treatment: a randomized controlled clinical trial of two initial aligning arch wires. Am J Orthod Dentofacial Orthop. 1992 Oct;102(4):373-81. doi: 10.1016/0889-5406(92)70054-e. PMID 1456222
- [Background] Lamberton JA, Oesterle LJ, Shellhart WC, Newman SM, Harrell RE, Tilliss T, Singh N, Carey CM. Comparison of pain perception during miniscrew placement in orthodontic patients with a visual analog scale survey between compound topical and needle-injected anesthetics: A crossover, prospective, randomized clinical trial. Am J Orthod Dentofacial Orthop. 2016 Jan;149(1):15-23. doi: 10.1016/j.ajodo.2015.08.013. PMID 26718373
- [Background] Steen Law SL, Southard KA, Law AS, Logan HL, Jakobsen JR. An evaluation of preoperative ibuprofen for treatment of pain associated with orthodontic separator placement. Am J Orthod Dentofacial Orthop. 2000 Dec;118(6):629-35. doi: 10.1067/mod.2000.110638. PMID 11113797
- [Background] Minor V, Marris CK, McGorray SP, Yezierski R, Fillingim R, Logan H, Wheeler TT. Effects of preoperative ibuprofen on pain after separator placement. Am J Orthod Dentofacial Orthop. 2009 Oct;136(4):510-7. doi: 10.1016/j.ajodo.2007.09.018. PMID 19815152
- [Background] Ngan P, Wilson S, Shanfeld J, Amini H. The effect of ibuprofen on the level of discomfort in patients undergoing orthodontic treatment. Am J Orthod Dentofacial Orthop. 1994 Jul;106(1):88-95. doi: 10.1016/S0889-5406(94)70025-7. PMID 8017354
- [Background] Ohnhaus EE, Adler R. Methodological problems in the measurement of pain: a comparison between the verbal rating scale and the visual analogue scale. Pain. 1975 Dec;1(4):379-384. doi: 10.1016/0304-3959(75)90075-5. PMID 800639
- [Background] Oliver RG, Knapman YM. Attitudes to orthodontic treatment. Br J Orthod. 1985 Oct;12(4):179-88. doi: 10.1179/bjo.12.4.179. PMID 3863673
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Ottoson D, Ekblom A, Hansson P. Vibratory stimulation for the relief of pain of dental origin. Pain. 1981 Feb;10(1):37-45. doi: 10.1016/0304-3959(81)90043-9. PMID 7232010
- [Background] Polat O, Karaman AI, Durmus E. Effects of preoperative ibuprofen and naproxen sodium on orthodontic pain. Angle Orthod. 2005 Sep;75(5):791-6. doi: 10.1043/0003-3219(2005)75[791:EOPIAN]2.0.CO;2. PMID 16279825
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Salmassian R, Oesterle LJ, Shellhart WC, Newman SM. Comparison of the efficacy of ibuprofen and acetaminophen in controlling pain after orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):516-21. doi: 10.1016/j.ajodo.2007.05.020. PMID 19361739
- [Background] Wilson S, Ngan P, Kess B. Time course of the discomfort in young patients undergoing orthodontic treatment. Pediatr Dent. 1989 Jun;11(2):107-10. PMID 2762180